CLINICAL TRIAL: NCT01450826
Title: A Randomized Open Label Phase II Trial of Aprepitant (Emend) in Combination With Ondansetron Compared to Standard 5HT3 Serotonin Antagonist (Ondansetron) in the Prevention of Acute and Delayed Chemotherapy Induced Nausea and Vomiting (CINV) in Glioma Patients Receiving a Temozolomide Based Regimen
Brief Title: Emend and Ondansetron Compared to Ondansetron Alone to Prevent CINV in Glioma Patients Receiving Temozolomide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Katy Peters (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Katy Peters, Assistant Professor, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00031206
Record Dates: First submitted 2011-10-10; First posted 2011-10-12 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: Nausea; Vomiting; Glioma
Keywords: Chemotherapy induced nausea and vomiting; CINV; Glioma; Temozolomide; Temodar; Aprepitant; Emend; Ondansetron; Zofran; Pro00031206; Affronti; Peters; Duke; Preston Robert Tisch Brain Tumor Center
MeSH Terms: conditions — Nausea; Vomiting; Glioma | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aprepitant+ondansetron (Active Comparator): On day 1, patients will receive a single oral dose of Aprepitant 125 mg p.o, 1 hour before first dose of the 5-day oral temozolomide regimen. This will be followed by Aprepitant 80 mg p.o. on days 2 -5 (1 hour prior to temozolomide). Additionally, On days 1-5, patients receive a single dose of Ondansetron 30 minutes before the receiving their prescribed dose of 5-day oral temozolomide.
  Interventions: Drug: aprepitant; Drug: ondansetron
- ondansetron (Active Comparator): On days 1-5, patients receive a single dose of Ondansetron 30 minutes before the receiving their prescribed dose of 5-day oral temozolomide.
  Interventions: Drug: ondansetron

INTERVENTIONS:
Drug: aprepitant — On day 1, eligible patients will receive a single oral dose of Aprepitant 125 mg p.o, 1 hour before first dose of the 5-day oral temozolomide regimen. This will be followed by Aprepitant 80 mg p.o. on days 2 -5 (1 hour prior to temozolomide).
  Other Names: Emend
  Arms: aprepitant+ondansetron
Drug: ondansetron — On Days 1-5, eligible patients will receive a single oral dose of Ondansetron, 30 minutes before first dose of the 5 -day oral temozolomide regimen.
  Other Names: Zofran

SUMMARY:
Patients diagnosed with malignant glioma who are receiving temozolomide will be accrued in this open label, phase 2, randomized single institution trial of aprepitant in combination with ondansetron versus ondansetron alone for the prevention of acute and delayed chemotherapy-induced nausea and vomiting (CINV). Sixty-eight (68) patients will be randomized to each arm of the study.

DETAILED DESCRIPTION:
Sixty-eight (68) patients will be randomized to each arm of the study. Patient randomization will be stratified by grade of tumor (1 or 2 versus 3 or 4) and the number of prior progressions (0 or 1 versus 2). Within each of the 4 strata defined by these factors, a permuted block randomization scheme will be used to assign patients to receive either aprepitant in combination with ondansetron or ondansetron alone.

Though the study is comparative, the goal of the study is to determine whether aprepitant is worthy of further investigation in this setting, and not to make definitive statements about the comparative effectiveness of ondansetron treatment with or without aprepitant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of glioma (either low or high grade) and be either chemotherapy naïve or non-naïve and scheduled to receive temozolomide-based +/- Bevacizumab- based chemotherapy. Patients with recurrent disease whose diagnostic pathology confirmed glioma (either low or high grade) will not need re-biopsy.
* Age ≥ 18 years
* ≤ 2 prior chemotherapeutic regimens
* Patient is scheduled to receive temozolomide at either 150 mg/m2 or 200mg/m2 by mouth for 5 days out of a 28 day cycle +/- bevacizumab.
* Study participation will occur during the first cycle of the 5 day temozolomide course.
* An interval of at least 6 weeks between prior surgical resection and study enrollment
* Karnofsky ≥ 60%.
* Hematocrit > 29%, absolute neutrophil count (ANC) > 1,000 cells/µl, platelets > 100,000 cells/µl
* Serum creatinine < 1.5 mg/dl, serum glutamic oxaloacetic transaminase (SGOT) and bilirubin < 1.5 times upper limit of normal
* For patients on oral corticosteroids, they must be stable clinically on corticosteroids or tapered off prior to starting the study drug. For patients taking dexamethasone, the dose should not exceed 8 mg qd (or 4 mg twice a day), if clinically stable, and the dose should not be escalated over entry dose level, if clinically possible. The patient's dose of dexamethasone will be evaluated by the PI, the patient's study physician, and/or the study pharmacist on a case by case basis for safety. All doses of oral corticosteroids will be reduced by 50% to avoid drug to drug interactions with Aprepitant, unless oral corticosteroids are at physiologic dose (e.g. dexamethasone 1 mg, prednisone 10 mg, or cortisone 30 mg). It is recommended that oral corticosteroid doses be escalated back to full dose on Day 7 (2 days after Aprepitant is discontinued) based on Aprepitant half-life pharmacokinetic data, and expert clinical opinion.
* Signed informed consent approved by the Institutional Review Board prior to patient entry
* If sexually active, patients will take contraceptive measures for the duration of protocol treatment and continue until one month after treatment. The efficacy of hormonal contraceptives during and for 28 days following the last dose of Aprepitant may be reduced. Alternative or back-up methods of contraception must be used.
* Approved rescue medication for the treatment of nausea and vomiting is permitted at the discretion of the investigator. The rescue antiemetics allowed will include: ondansetron, granisetron and lorazepam.

Exclusion Criteria:

* Pregnant or breast-feeding (While both aprepitant and ondansetron are classified as Category B drugs, an eligibility criteria for this study is that the patient be scheduled to receive a temozolomide-based chemotherapy regimen +/- bevacizumab, which are Category D and C drugs respectively. Therefore, while not considered necessary for the administration of the current study drugs, a pregnancy test should be a part of normal clinical care for the patients in this study, if the patient is determined to be of child-bearing potential.)
* No prior nitrosourea (e.g. lomustine, carmustine)
* Inability or unwillingness to understand or cooperate with study procedures
* Concurrent administration of CYP3A4 enzyme-inducing anti-epileptic drugs (EIAEDs) including phenytoin, phenobarbitol, carbamazepine, oxcarbazepine or primidone
* Prohibited medications: Patients taking CYP3A4 enzyme inducers and moderate or strong inhibitors will be excluded from this trial.
* Received any drug with potential anti-emetic effect within 24 hours prior to the start of study-designated chemotherapeutic agent: HT3 receptor or substance P/neurokinin 1(NK1) receptor antagonists; Dopamine receptor antagonists (metoclopramide); Phenothiazine anti-emetics (prochlorperazine, thiethylperazine and perphenazine); Diphenhydramine, scopolamine, chlorpheniramine maleate, trimethobenzamide; Haloperidol, droperidol, tetrahydrocannabinol, or nabilone
* Any vomiting, retching or NCI Common Toxicity Criteria v.4.0 grade 2-4 nausea 24 hours preceding chemotherapy
* Ongoing vomiting from any organic etiology
* Will receive radiotherapy of cranium within one week prior to or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-06-24 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Affronti, DNP, RN, MHSc, ANP, Principal Investigator — Duke University; Katherine B Peters, MD, PhD, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center — https://tischbraintumorcenter.duke.edu/
- See also: Duke Cancer Institute — http://www.dukecancerinstitute.org/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aprepitant+Ondansetron | Ondansetron
Started | 70 | 66
Completed | 70 | 66
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant+Ondansetron | Ondansetron | Total
Number analyzed (Participants) | 70 | 66 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.96 (14.25) | 55.03 (12.17) | 53.96 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 24 | 53
  Male | 41 | 42 | 83
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving Complete Control (CC)
Description: Complete control (CC): study days 1-7 (acute and delayed CINV) the proportion of patients achieving complete control (CC); defined as no emetic episode, no need for rescue medication during days 1-7; number of emetic episodes daily; time to first emetic episode; as captured by the MAT (MASCC Antiemesis Tool)/Osoba survey (MASCC refers to Multinational Association for Supportive Care in Cancer™). Severity of nausea and other toxicities measured daily by the NCI Common Toxicity Criteria (version 4.0).
Time Frame: 7 days
Population: Intent to treat
Measure: Number; unit: proportion of patients
Arm/Group | Aprepitant+Ondansetron | Ondansetron
Number analyzed (Participants) | 70 | 66
proportion of patients | 0.59 | 0.55

2. Secondary Outcome: Proportion of Patients Achieving an Acute and Delayed Complete Response (CR)
Description: CR is the proportion of patients with no emetic episode and no rescue medication. (1) Assessed from the beginning of study day 1, CR is defined for acute CINV as no emetic episode and no use of rescue anti-nausea medication during the first 24 hours following chemotherapy administration. An emetic episode is defined as one episode of vomiting or a sequence of episodes in very close succession not relieved by a period of relaxation of at least 1 min, any number of unproductive emetic episodes (retches) in any given 5 minute period, or an episode of retching lasting <5 minutes combined with vomiting not relieved by a period of relaxation of at least 1 minute; (2) Complete response (CR) on study days 2-7 (delayed CINV) is defined as the proportion of patients achieving a CR during the delayed time period. The data will be captured by the validated ultinational Association of Supportive Care in Cancer (MASCC) Anti-emesis Tool (MAT)/Osoba survey.
Time Frame: 7 days
Population: Intent to treat
Measure: Number; unit: proportion of patients
Arm/Group | Aprepitant+Ondansetron | Ondansetron
Number analyzed (Participants) | 70 | 66
proportion of patients
  Acute CINV CR | 0.97 | 0.88
  Delayed CINV CR | 0.59 | 0.58

3. Secondary Outcome: Patient's Global Satisfaction With the Antiemetic Regimen
Description: Patients' global satisfaction with the antiemetic regimen is measured using the Osoba survey, which was administered on days 1-7. This survey asks patients "In the past 24 hours, did vomiting or dry heaves a) interfere with your appetite, b) affect your sleep, c) interfere with your physical activities, d) interfere with your social life, and e) interfere with your enjoyment of life?" Patients responded on a scale of 1-4 ranging from 'Not at all' to 'Very much.' Global satisfaction was defined as responding 'Not at all' for all questions related to vomiting/retching for each study day. The proportion of patients responding 'Not at all' for all Osoba vomiting/retching questions over the study period is reported.
Time Frame: 7 days
Population: 2 patients in the Aprepitant + Ondansetron arm and 4 patients in the Ondansetron arm did not have adequate survey data for this analysis
Measure: Number; unit: proportion of patients
Arm/Group | Aprepitant+Ondansetron | Ondansetron
Number analyzed (Participants) | 68 | 62
proportion of patients | 0.87 | 0.81

4. Secondary Outcome: Time to Treatment Failure
Description: Median time in days to first emetic episode or first need of rescue medication, whichever occurred first as measured by the MAT/Osoba survey, among those patients experiencing an emetic episode or need of rescue medication
Time Frame: 7 days
Population: This analysis only includes those patients no achieving complete control (no emetic episode or need for rescue medication throughout the 7-day study period).
Measure: Median (Full Range); unit: days
Arm/Group | Aprepitant+Ondansetron | Ondansetron
Number analyzed (Participants) | 29 | 30
days | 5 [1 to 7] | 4 [1 to 7]

ADVERSE EVENTS:
Time Frame: 30 days
Groups:
- Ondansetron Alone: On days 1-5, patients receive a single dose of Ondansetron 30 minutes before the receiving their prescribed dose of 5-day oral temozolomide.
  Ondansetron: On Days 1-5, eligible patients will receive a single oral dose of Ondansetron, 30 minutes before first dose of the 5 -day oral temozolomide regimen.
Arm/Group | Aprepitant+Ondansetron | Ondansetron Alone
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/66
Serious Adverse Events (participants affected / at risk) | 1/70 | 3/66
Other Adverse Events (participants affected / at risk) | 57/70 | 51/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant+Ondansetron (N=70) | Ondansetron Alone (N=66)
Dysphasia (Nervous system disorders) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: R HEMIPLEGIA DUE TO DISEASE PROGRESSION (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aprepitant+Ondansetron (N=70) | Ondansetron Alone (N=66)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 9 | 7
Diarrhea (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify: LIKELY VIRUS: DIARRHEA, FATIGUE, LOW GRADE FEVER (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 37 | 37
Vomiting (Gastrointestinal disorders) | 7 | 5
Chills (General disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Fatigue (General disorders) | 20 | 13
Fever (General disorders) | 1 | 2
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 0
Injury, poisoning and procedural complications - Other, specify: LACERATION REQUIRING STITCHES (Injury, poisoning and procedural complications) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
White blood cell decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 6 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Dysphasia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 6 | 5
Nervous system disorders - Other, specify: DIFFICULTY WALKING AND GETTING UP FROM SITTING POSITION (Nervous system disorders) | 1 | 0
Nervous system disorders - Other, specify: R FACIAL DROOP DUE TO DISEASE PROGRESSION (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 3 | 4
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2
Skin and subcutaneous tissue disorders - Other, specify: RASH TO CHEST; TEMO;UNRELATED TO EMEND (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify: RASH; EMEND (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-20): https://cdn.clinicaltrials.gov/large-docs/26/NCT01450826/Prot_SAP_000.pdf